CLINICAL TRIAL: NCT05865288
Title: The Moderating Role of Baseline Oxytocin on Its Psychotherapy-facilitating Effects Among Patients With Eating Disorders
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHA-0007-23
Record Dates: First submitted 2023-03-21; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Eating Disorders
Keywords: Oxytocin; eating disorders; cognitive rigidity
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): 24IU (12IU*2) of Oxytocin, Sorbitol, Benzyl, alcohol glycerol, distilled water.
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator): 24IU (12IU*2) of Sorbitol, Benzyl, alcohol glycerol, distilled water.
  Interventions: Drug: Oxytocin nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal OT will be performed using a spray containing 24IU (12IU administered to each nostril), sorbitol, benzyl, alcohol glycerol, distilled water. Dosage and administration method was determined by standard OT studies instructions and guidelines. The substance will be prepared immediately after randomization by an external preparation and delivered and stored until administration under required conditions. The nasal spray will be self administered, with the nursing staff supervising for proper administration of substance, after training and guiding the patient, and for supervision of side effects.

SUMMARY:
Introduction: Oxytocin (OT) is a nine-amino acid neuropeptide known to play a vital part in social behaviors and has also been found to be involved the social manifestations of mental illnesses, such as social manifestations and social cognition. it has been suggested that OT administration may serve as an add-on treatment for individuals with mental illnesses.

One group of patients affected by social are patients with eating disorders (EDs). Studies of OT administration among individuals with EDs have shown an inconsistent pattern of findings, which might be associated with the differential baseline level of OT dysregulation. Thus OT dosing needs to be optimized, while considering patients baseline OT levels prior to administration. Patients with ED are also known to have lower OT levels at baseline. It is possible that OT's administration will affect interpersonal behavior through the increase of lowered OT levels, thus leading to overall improvement of ED symptoms.

This study aims to examine the effects of OT administration among patients with EDs, while focusing on baseline OT levels and interpersonal abilities as potential moderators and/or mediators of its effects. The research addresses the following questions: (1) is OT administration associated with increased therapeutic gains among patients with ED? (2) what are the moderators and mediators of these effects, and specifically, do baseline levels of OT and baseline interpersonal abilities moderate these effects? (3) what is the mechanism underlying OT's therapeutic effects, and specifically do changes in interpersonal abilities and changes in OT levels serve a mediating role? Methods: This study aims to assess the differential effect of OT administration among patients with varying levels of baseline saliva OT and to explore the effects of optimizing frequency and dosage of administration of OT, based on baseline characteristics.

Participants: Female and male Individuals (N=90) with verified diagnosis of EDs, age 16 and above, will participate in at least four weeks of treatment at the EDs unit. Subjects will be recruited at the Teradion Eating Disorder Clinic, an outpatient unit in North Israel.

Procedure: Patients and caregivers will sign an informed consent form. Baseline saliva OT will be measured four times during consecutive days. At week 1 patients will be assessed for general distress, ED symptoms, cognitive rigidity, interpersonal abilities, as well as patients and therapists reported working alliance. At week 2 patients will be randomized at a ratio of 2:1 with 60 patients receiving OT and 30 receiving placebo. Patients will receive 24 IU of OT or placebo, once a week, prior to therapy sessions, for a period of 4 weeks. During these weeks (2-5), they will be assessed for levels of OT, general distress, interpersonal abilities, working alliance and cognitive rigidity. All measurements will be performed finally at week 6.

Novelty: This study is the first to assess the effectiveness of OT as an add-on for patients with EDs, during clinical treatment, as well as to explore modulators such as baseline OT levels, and mediators such as social abilities and cognitive rigidity, on the overall improvement of ED patients in therapy.

DETAILED DESCRIPTION:
Introduction: Oxytocin (OT) is a nine-amino acid neuropeptide known to play a vital part in social behaviors and has also been found to be involved the social manifestations of mental illnesses. Based on correlations found between OT levels and psychiatric symptoms, such as social manifestations, trust and social cognition. It has been suggested that OT administration may serve as an add-on treatment for individuals with mental illnesses.

One group of patients known to be profoundly affected by deficits in social bonding, social cognition and trust are patients with eating disorders (EDs). Studies assessing the potential beneficial effect of OT administration among individuals with EDs have shown an inconsistent pattern of findings, which might be associated with the differential baseline level of OT dysregulation.

It has been suggested that OT dosing might need to be optimized, possibly while considering patients baseline OT levels prior to administration, as well as other possible clinical, personality and demographic characteristics. OT's effects are largely associated with social and interpersonal aspects and cognitive aspects of human behavior, therefore serving as a potential mechanism to explain its beneficial effects in patients with EDs, through the modulation of social and cognitive routes. Patients with ED, who are characterized by such social deficits, lack of trust in caregivers, and cognitive rigidity might have a significant beneficial effect from OT administration, as these patients are also known to have lower OT levels at baseline. It is is possible that OT's administration will affect interpersonal behavior through the increase of these lowered OT levels, thus leading to overall improvement of ED symptoms.

In this study investigators aim to examine the effects of OT administration among patients with eating disorders (EDs), while focusing on baseline OT levels and interpersonal abilities as potential moderators and/or mediators of its effects. The research is designed to address the following research questions: (1) Is OT administration associated with increased therapeutic gains among patients with ED? (2) What are the moderators and mediators of these effects, and specifically, do baseline levels of OT and baseline interpersonal abilities moderate these effects? (3) What is the mechanism underlying OT's therapeutic effects, and specifically do changes in interpersonal abilities and changes in OT levels serve a mediating role?

Based on the literature review, the following research hypotheses were made:

(I) Oxytocin administration will have an overall small to moderate beneficial effect to patients with ED.

(II) Baseline levels of OT will moderate this effect, such that patients with lower levels of OT will produce better symptomatic outcomes following OT administration compared to patients with high OT levels.

(III) Patients with low baseline OT levels, as well as low social abilities, will benefit the most from OT administration.

(IV) Changes in social abilities and in OT levels will serve as mediators to OT's effects.

Furthermore, cognitive rigidity and therapists and patients working alliance will be measured for exploratory future analyses.

Methods:

This study is designed as a proof-of-concept RCT, aimed to assess the differential effect of OT administration among patients with varying levels of baseline saliva OT. This study serves as the infrastructure for the second phase of the study, aimed to explore the effects of optimizing frequency and dosage of administration of OT, based on baseline characteristics.

Participants:

Female and male Individuals (N=90) with EDs will be recruited. Inclusion criteria will include: (1) aged 16 and above, (2) verified diagnosis of ED, (3) at least four weeks are expected in treatment at the EDs unit. Exclusion criteria will include: (1) no ongoing medical care (patients leaving treatment during the study will be excluded), (2) immediate suicidal or violent risk, (3) inability to complete self-report measures for any reason, (4) pregnancy.

Subjects will be recruited at the Teradion Mental Health -Eating Disorder Clinic, an outpatient unit located in the northern area of Israel. The unit provides treatment to patients with eating disorders (mainly AN, BN and BED), and includes a multi-professional staff of psychiatrists, psychologists, social workers, and dietitians.

Procedure:

Patients agreeing to participate will sign an informed consent form. Patients under the age of 18 will participate only if both parents and the patient signed informed consent. After signature has been obtained, baseline saliva OT will be measured four times during four consecutive days. During this phase (week 1), patients will be assessed for general distress, ED symptoms, cognitive rigidity, interpersonal abilities, as well as patients and therapists reported working alliance. After baseline measurements are complete (week 2), patients will be randomized at a ratio of 2:1 to receive OT or placebo, with 60 patients receiving OT and 30 receiving placebo. Randomization will be performed by a staff member blind to the study objectives. Administration of OT will be performed by a nurse blind to the study objectives. Patients will receive 24 IU of OT or placebo, once a week, prior to therapy sessions, for a period of 4 weeks. During these weeks (week 2-5), they will be assessed for levels of OT, general distress, interpersonal abilities, patients and therapists working alliance and cognitive rigidity. A second wave of OT measurement will be performed in week 6.

Measures:

The Hopkins symptoms checklist -short form : The HSCL-11 is a brief version of the SCL-90-R and includes 11 items assessing general symptomatic distress through self-report. The HSCL-11 was previously found suitable for detecting weekly changes in symptom severity during the course of treatment in major depression disorder patients. In order assess changes in general distress, as manifested by anxiety and depression symptoms the HSCL-11 will be delivered at baseline, and on a weekly basis.

The Eating Disorder Examination Questionnaire (EDEQ). The EDEQ (v 6.0) is a 28-item self-reported questionnaire, adapted from the semi-structured interview Eating Disorder Examination (EDE) and designed to assess the range and severity of features associated with a diagnosis of eating disorder using 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and a global score. The EDEQ will be completed at baseline and once weekly.

The Detail and Flexibility Questionnaire (DFlex). The DFlex is a 24-item self-report scale aimed to measure two aspects of neurocognitive functioning: cognitive rigidity (difficulty with set shifting/flexibility) and attention to details. The 24 items are rated on an agreement/disagreement scale ranging from 1 to 6, with higher scores indicating higher cognitive rigidity and lower scores indicating higher flexibility. The DFlex will be completed at baseline and once weekly.

The Inventory of Interpersonal Problems (IIP short version). The IIP short version is a 32-item self-report measure of interpersonal distress. This self-report inventory asks participants to rate a variety of interpersonal problems that may cause distress. The items are divided into two groups: (1) interpersonal inadequacies or inhibitions (20 items), (2) excesses or compulsions (12 items). The items in the first group all start with the phrase "It is hard for me to…", whereas the items in the second group involve the phrase "too much". Participants rate each item on a scale from 0 to 4 on how much difficulty/distress they feel regarding the item.

The Working Alliance Inventory - Short Revised (WAI - SR). A 12-item self-report questionnaire aimed to evaluate patient-therapist working alliance through three aspects: agreement on therapy goals, agreement on therapeutic tasks and patient-therapist positive emotional bond. It is rated on a 6-point scale ranging from not at all (1) to very much (6). The questionnaire has two versions: one assessing the alliance from the patient's point of view and the other assessing it from the therapist's point of view (see Appendix D). Both patients and therapists will complete the WAI-12 every week during administration.

Measurement of OT Oxytocin baseline levels will be measured in participants' saliva via test tubes. Saliva will be measured four times, preferably in early morning before food consumption, and an average baseline will be calculated.

Administration of OT Intranasal OT will be performed using a spray containing 24IU (12IU administered to each nostril).Control-placebo group will be administered using the same spray, containing the same components but the OT.

Statistical strategy Multilevel models will be performed to assess the effects of OT administration in patients receiving OT versus those receiving placebo. The moderating effect of baseline OT levels, social abilities, and cognitive rigidity at baseline will be assessed by adding these variables as second level interaction terms in MLM models. To identify patients which are most likely to profit from OT administration, group and baseline characteristics, including mean baseline OT levels, will be entered as predictors in Elastic Net Penalized Logistic Regressions (ELNET) to assess predictive factors to optimal reliable clinical change. The mediating effects of changes in working alliance, social abilities, and cognitive rigidity levels will be tested by the Hayes PROCESS macro.

Ethical considerations

This research will be performed in accordance with ethical principles of Helsinki WMA Declaration. Patients and therapists will sign informed consent forms before participating in any study related procedures. Previous studies have shown that the IN-OT side-effects are very low. Minor side effects reported by 5-6% of the patients included an increase in calmness\euphoric sensation, light headedness, dry mouth, restlessness, nervousness and headache, and a sense of stimulation in the nostrils and dryness in mouth were reported by 3% of participants.

Information safety Clinical data obtained from the facilities of Teradion MH-EDC, and the participants' blinded data will be collected and stored in safely guarded computers of Clalit Health Services, or a locked closet in the Clinic for 7 years, and then will be shredded.

The Novelty of the study is in being is the first to assess the effectiveness of OT as an add-on for patients with EDs, during clinical treatment, as opposed to a single given dose, and to further explore modulators such as baseline OT levels, and mediators such as social abilities and cognitive rigidity, on the overall improvement of ED patients in therapy.

ELIGIBILITY:
Patients Inclusion Criteria:

* verified diagnosis of ED
* at least four weeks of treatment at the EDs unit

Patients Exclusion Criteria:

* no ongoing medical care
* immediate suicidal or violent risk
* inability to complete self-report measures for any reason
* pregnancy according to self report

Therapist Inclusion Criteria:

* psychologists, psychiatrists, social workers, Dieticians, and art therapist in different stages of seniority and training.

Therapist Exclusion Criteria:

* pregnancy according to self-report.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
eating disorder symptoms | 6 weeks
  as measured by the EDEQ -Eating disorder examination questionnaire, a 28-item self-reported questionnaire, using 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and a global score (Fairburn & Beglin, 1994).

SECONDARY OUTCOMES:
general symptomatic distress | 6 weeks
  as measured by HSCL - The Hopkins symptoms checklist -short form (Lutz, Tholen, Schürch, & Berking, 2006).
cognitive rigidity | 6 weeks
  as measured by DFlex - Detail and Flexibility Questionnaire Roberts et al., 2011).
social deficits | 6 weeks
  as measured by the IIP short version - Inventory of Interpersonal Problems (Gurtman, 1996)
working alliance | 6 weeks
  as measured by WAI-SR - The Working Alliance Inventory - Short Revised (Hatcher & Gillapsy, 2006).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Shalvata Mental health Center, Hod HaSharon
  - Eating Disorder Clinic, Teradion, Misgav Regional Council